CLINICAL TRIAL: NCT05608733
Title: Continuous Sciatic Nerve Block vs Epidural Analgesia in Lower Limb Amputation for Prevention of Acute Postoperative Pain and Phantom Limb Pain: A Triple-blind Randomized Controlled Non-inferiority Clinical Trial.
Brief Title: Continuous Sciatic Nerve Block vs Epidural Analgesia in Lower Limb Amputation for Postoperative Pain
Acronym: Ampupain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IN-47-2021
Record Dates: First submitted 2022-03-09; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-03

CONDITIONS: Phantom Limb Pain; Pain, Chronic
MeSH Terms: conditions — Phantom Limb; Chronic Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural catheter (Experimental): Epidural catheter infusion of bupivacaine 0.1% (4-6 cc/h) at level L3-L4
  Interventions: Drug: Epidural catheter
- Continuous sciatic nerve block (Active Comparator): Continuous sciatic catheter infusion of bupivacaine 0.1% (6-10 cc/h)
  Interventions: Drug: Continuous sciatic nerve block

INTERVENTIONS:
Drug: Epidural catheter — Bony landmarks and the space between the lower lumbar vertebrae are identified. Subsequently, infiltration of the skin and subcutaneous cellular tissue with local anesthetic (Lidocaine 2% without epinephrine) is performed at the site to be punctured. A 17G Tuohy needle is inserted 2-4 cm through the skin, then the mandrel is removed, the low-resistance syringe is connected, and the loss of resistance is checked using the air or liquid technique, depending on the preference of the anesthesiologist. . Appreciating the loss of resistance in the embolus, the mandrel is then withdrawn and the epidural catheter is advanced to leave it an additional 5 cm inside the epidural space.
  Other Names: Epidural Analgesia
  Arms: Epidural catheter
Drug: Continuous sciatic nerve block — The patient is placed in the prone or supine position with the limb to be blocked flexed at 90°. Using a high-frequency linear transducer and using sterile technique, the popliteal sciatic nerve is identified in an axial axis. A 17G Tuohy needle is inserted plane and medial. Saline solution (5 ml) is applied to open the perineural space. Adequate hydrodissection and donut sign in the nerve are observed..A perineural catheter is then advanced 5 cm beyond the tip of the needle. The catheter is fixed with stitches and a transparent sterile dressing is placed.
  Other Names: Periferical continuous block
  Arms: Continuous sciatic nerve block

SUMMARY:
Controlled clinical trial of two parallel groups, with random assignment 1:1, non-inferiority, blinded for the patient, for who administers the intervention and for who analyzes the data. 112 participants

DETAILED DESCRIPTION:
Controlled clinical trial of two parallel groups, with random assignment 1:1, non-inferiority, blinded for the patient, for who administers the intervention and for who analyzes the data. 112 participants Outcomes: Primary: Numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain) was used for pain assessments daily for 15 days and subsequently monthly until completing 3 months. Co-primary: Assessment of symptomatology related to phantom limb pain daily for 15 days POP and subsequently monthly until completing 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Being scheduled for above or below knee amputation or for bone remodeling of lower limb amputees
3. Acceptance of continuous regional analgesic technique as part of their multimodal analgesia

Exclusion Criteria:

1. Traumatic cause of amputation
2. Allergy to local anesthetics
3. Contraindication for epidural technique or continuous blocks
4. Stage 5 kidney disease
5. Concomitant use of aspirin and clopidogrel
6. Pregnancy status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Posoperative Pain | 3 months
  Pain score according to the daily NRS scale (Numeric Pain Rating Scale), Numeric Pain Rating Scale, for 15 days POP and subsequently monthly until completing 3 months. is scores from 0 to 10, 10 being the worst value.
Phantom Limp Pain | 3 months
  For this qualitative dichotomous outcome, you will ask about symptomatology referring to phantom limb pain for 15 days POP and subsequently monthly until completing 3 months, It will be qualified as positive if it presents any neuropathic symptom.

SECONDARY OUTCOMES:
Phantom Limp Pain first Year | 1 year
  Presence of phantom limb pain on a monthly basis until completing 12 month, The patient will be asked about the appearance of any painful sensation described as stabbing, shooting, electric shock, dull, tight pain and/or cramp in the anatomical site where the amputated limb would be, evaluating the presence or absence of the same (s). This will be questioned every day for 15 POPs days and monthly follow-up will continue via telephone until completing 3 months.
Opioid Consumption | 36 hours
  the total consumption in mg of morphine or its equivalent at 12, 24 and 36 h POP will be evaluated.
Incidence of nausea and vomiting POP | 36 hours
  Incidence of nausea and vomiting POP in each group: the appearance of nausea or vomiting at 12, 24 and 36 h POP will be asked.
Incidence of adverse effects | 1 year
  any appearance of hematoma, hypotension (defined as SBP less than 90 mmHg or a 30% decrease in baseline MAP) or bradycardia (HR less than 60 bpm) is defined.
Days of hospital stay | during the time of hospitalization, on average 10 days
  Days of hospital stay through study completion
Mortality | 1 year
  Mortality in the first Year

OTHER OUTCOMES:
Posoperative Satisfaction | 36 hours
  Postoperative satisfaction measured with the EVAN LR scale (evaluation of local anesthetic satisfaction).
  It consists of a self-reported scale that measures satisfaction in the postoperative period of patients undergoing regional anesthesia in different surgical models (51), with an evaluation of 19 items structured in a global index and five unweighted dimensions, each of which covers some aspects such as Attention (4 items), Information (5 items), Discomfort (4 items), Waiting (2 items) and Pain (4 items).
  has a score for questions between 20 and 100 points, the lower the score, the lower satisfaction by dimension

CONTACTS AND LOCATIONS:
Overall Officials: Mario Zamudio, Prof, Study Director — IPS universitaria
Locations (1):
- Antioquia´s University, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No
public bases of data

REFERENCES:
- [Background] Edgley C, Hogg M, De Silva A, Braat S, Bucknill A, Leslie K. Severe acute pain and persistent post-surgical pain in orthopaedic trauma patients: a cohort study. Br J Anaesth. 2019 Sep;123(3):350-359. doi: 10.1016/j.bja.2019.05.030. Epub 2019 Jun 24. PMID 31248645
- [Background] De Jong R, Shysh AJ. Development of a Multimodal Analgesia Protocol for Perioperative Acute Pain Management for Lower Limb Amputation. Pain Res Manag. 2018 Jun 3;2018:5237040. doi: 10.1155/2018/5237040. eCollection 2018. PMID 29973967
- [Background] Gehling M, Tryba M. [Prophylaxis of phantom pain: is regional analgesia ineffective?]. Schmerz. 2003 Jan;17(1):11-9. doi: 10.1007/s00482-002-0198-2. German. PMID 12579385